CLINICAL TRIAL: NCT03973879
Title: A Phase 1b/2 Trial of PVSRIPO in Combination With Atezolizumab in Recurrent WHO Grade IV Malignant Glioma
Brief Title: Combination of PVSRIPO and Atezolizumab for Adults With Recurrent Malignant Glioma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Re-submission Planned
Sponsor: Darell Bigner (Other)
Collaborators: Istari Oncology, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Darell Bigner, Sponsor-Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100677
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Malignant Glioma
Keywords: PVSRIPO; Atezolizumab; Glioblastoma; Glioma; Bigner; Randazzo; Brain tumor; Duke; Istari; Pro00100677; Genentech
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PVSRIPO + Atezolizumab (Experimental): Single PVSRIPO infusion at a dose of 5x10^7 tissue culture infected dose (TCID50). Atezolizumab infusions at a dose of 1200 mg every three weeks for up to two years.
  Interventions: Biological: PVSRIPO; Drug: Atezolizumab

INTERVENTIONS:
Biological: PVSRIPO — Oncolytic polio/rhinovirus recombinant
Drug: Atezolizumab — Antibody
  Other Names: Tecentriq

SUMMARY:
This study evaluates the safety of PVSRIPO treatment in combination with Atezolizumab in patients with WHO grade IV malignant glioma. All patients will receive a single PVSRIPO infusion followed by atezolizumab infusions every three weeks for up to two years.

DETAILED DESCRIPTION:
The purpose of this phase1b/2 study of atezolizumab in combination with oncolytic polio/rhinovirus recombinant (PVSRIPO) in patients with recurrent World Health Organization (WHO) grade IV malignant glioma is to assess the safety of the combination of PVSRIPO + atezolizumab, as well as describe the survival of patients receiving this novel therapy combination. Patients will receive an intratumoral infusion of PVSRIPO followed by atezolizumab treatment with possible surgical resection after the first atezolizumab treatment at the discretion of the treating neurosurgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a recurrent supratentorial WHO grade IV malignant glioma based on imaging studies with measurable disease (≥ 1 cm and ≤ 5.5 cm of contrast-enhancing tumor). Prior histopathology consistent with a WHO grade IV malignant glioma confirmed by the study pathologist, Roger McLendon, or his designate. Assuming patient meets all other criteria, the treating neurosurgeon must confirm placement of infusion catheter tip can occur ≥ 1cm from ventricles and that procedures can be completed per their medical judgement and in keeping with the protocol, when considering individual lesion characteristics including location relative to eloquent brain function.
* Patient or partner(s) meets one of the following criteria:

  1. Non-childbearing potential (i.e. not sexually active, physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile, or any male who has had a vasectomy). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Postmenopausal for purposes of this study is defined as 1 year without menses.; or
  2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g. birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g. a condom or diaphragm) used with spermicide.
* Age ≥ 18 years of age at the time of entry into the study
* Karnofsky Performance Score (KPS) ≥ 70%
* Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to biopsy
* Total bilirubin, serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), alkaline phosphatase ≤ 2.5 x normal prior to biopsy
* Neutrophil count ≥ 1000 prior to biopsy
* Hemoglobin ≥ 9 prior to biopsy
* Platelet count ≥ 100,000/µl unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 120,000/µl is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion
* Creatinine ≤ 1.2 x normal range prior to biopsy
* Positive serum anti-poliovirus titer prior to biopsy
* The patient must have received a boost immunization with trivalent inactivated IPOL™ (Sanofi-Pasteur) at least 1 week, but less than 6 weeks, prior to administration of the study agent
* At the time of biopsy, prior to administration of virus, the presence of recurrent tumor must be confirmed by histopathological analysis
* A signed informed consent form approved by the Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study
* Able to undergo brain MRI with and without contrast

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
* Patients with severe, active co-morbidity, defined as follow:

  1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
  2. Patients with known immunosuppressive disease or known human immunodeficiency virus infection
  3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
  4. Patients with known lung (forced expiratory volume in the first second of expiration (FEV1) < 50%) disease or uncontrolled diabetes mellitus
  5. Patients with albumin allergy
  6. Patients with gadolinium allergy
* Patients with a previous history of neurological complications due to PV infection
* Patients who have not recovered from the toxic effects of prior chemo- and/or radiation therapy. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used
* Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks) or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from side effects of such therapy
* Patients may not have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy
* Patients may not be less than 12 weeks from radiation therapy of the brain, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation
* Patients who have not completed all standard of care treatments for recurrent glioma, including surgical procedure and radiation therapy (at least 59 Gy)

  1. If the MGMT promoter in their tumor is known to be unmethylated, patients are not mandated to have received chemotherapy prior to participating in this trial
  2. If the MGMT promoter in their tumor is known to be methylated or the MGMT promoter methylation status is unknown at time of screening, patients must have received at least one chemotherapy regimen prior to participating in this trial
* Patients with neoplastic lesions in the brainstem, cerebellum, or spinal cord; radiological evidence of active (growing) disease (active multifocal disease); tumors with contrast-enhancing tumor component crossing the midline (crossing the corpus callosum); extensive subependymal disease (tumor touching subependymal space is allowed); or extensive leptomeningeal disease (tumor touching leptomeninges is allowed).
* Patients with undetectable anti-tetanus toxoid immunoglobulin G (IgG)
* Patients with known history of agammaglobulinemia
* Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to the first atezolizumab infusion
* Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups)
* Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Patients with a known history of hypersensitivity to atezolizumab, or any components of atezolizumab
* Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months

NOTE: If a patient is treated for an unrelated malignancy other than the exceptions noted within the past 3 years, a letter from their treating oncologist for the unrelated malignancy must be on file confirming that said unrelated malignancy does not require current active treatment (prophylactic like tamoxifen OK) and that the patient is stable with low risk of recurrence/death within 3 years from this other malignancy (i.e., disease is stable). If this letter is not on file, a consult with the Sponsor's medical designee is required prior to submitting the patient for consideration of enrollment in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Number of unacceptable adverse events | 14 days after first atezolizumab treatment
  Any Grade 3 or any Grade 4 toxicity that is not reversible within 2 weeks, or any life-threatening event, or treatment-related death.
Proportion of patients alive | 24 months after PVSRIPO infusion
  Proportion of patients alive at 24 months after PVSRIPO infusion

CONTACTS AND LOCATIONS:
Overall Officials: Darell D Bigner, MD, PhD, Study Director — Istari Oncology, Inc.; Dina M Randazzo, DO, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — https://www.dukehealth.org/clinical-trials